CLINICAL TRIAL: NCT04825262
Title: Efficacy of Achieving Early Target Trough Levels of Tacrolimus Using CYP3A5 Guided Dosing Versus Weight-based Dosing in a Multi-ethnic Population of Kidney Transplant Recipients in Singapore
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2019/2599
Record Dates: First submitted 2021-03-26; First posted 2021-04-01 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Kidney Transplant Rejection; Kidney Transplant; Complications
Keywords: kidney transplant; tacrolimus; CYP3A5; Pharmacogenomics
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Intervention Model Description: Single interventional group with historical control group
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention genotyping group (Experimental): Patients who are scheduled to receive renal transplant from a living donor between January 2021 to January 2023. They will be assigned to receive the initial CYP3A5 genotype-based tacrolimus (FK) dose as determined by their CYP3A5 genotype.
  CYP3A5 expresser (extensive or intermediate metabolizer) - 0.20mg/kg CYP3A5 non-expresser (poor metabolizer) - 0.15mg/kg
  The starting dose of the intervention arm will be reviewed for every 10 patients recruited based on the drug levels achieved.
  Interventions: Drug: Tacrolimus
- Historical Control Group (No Intervention): Patients who received renal transplant from a living donor between January 2016 - December 2020 and received standard weight-based dosing of tacrolimus

INTERVENTIONS:
Drug: Tacrolimus — Starting dose based on CYP3A5 genotype
  Arms: Intervention genotyping group

SUMMARY:
The investigators hypothesise that the adaptation of CYP3A5 genotype-based Tacrolimus (FK) dosing will lead to earlier FK target achievement and consequently, better clinical outcome after kidney transplantation (RTx).

This study aims to shed light on the possible impact of CYP3A genotype-based FK dosing on FK target achievement and clinical outcome after RTx in a multi-ethnic population where current evidence is lacking. This data would be helpful to the physicians so that by knowing the genotype of the patient before undergoing transplantation, practitioners would be able to decide on the starting dose of FK so as to avoid low trough levels and risk of acute rejection or high trough levels and risk of nephrotoxicity.

DETAILED DESCRIPTION:
Tacrolimus (FK) remains the cornerstone of maintenance immunosuppressants after renal transplantation. However, it is characterised by narrow therapeutic index and large inter-individual variability in its pharmacokinetics, particularly in the dose required to reach target trough blood concentrations. Among several factors investigated for their possible influence on tacrolimus pharmacokinetics, polymorphisms in genes coding for biotransformation enzymes (cytochrome P450 (CYP) isoenzymes 3A4 and 3A5) have received much attention. Exposure to FK correlates with the cytochrome P450 (CYP) 3A4 and CYP3A5 which are polymorphically expressed. This is in part explained by the presence of single-nucleotide polymorphisms (SNPs) in the CYP3A5 and CYP3A4 genes.

To date, renal transplant (RTx) recipients receive standard weight-based dosing of FK and therapeutic drug monitoring is employed for subsequent dose adjustment to ensure target FK concentration is attained. However, the current weight-based dosing strategies to guide the initial FK dosing have been poorly predictive of the actual FK dose required to attain therapeutic FK level. With the increased possibility of sub-therapeutic FK level during the early phase post renal transplantation, it puts them at a higher risk of developing acute rejection.

There has been increasing evidence to suggest the implementation of pre-transplantation genotyping to guide the initial FK dose to achieve target FK concentrations as quickly as possible. On the contrary, there are a few studies that report contradictory results of genotype-guided FK dosing as being useful in attainment of target therapeutic levels.

Given the differences in CYP3A5 genotype prevalence among races and the controversy in clinical benefits of such a pro-active dosage strategy, the impact of CYP3A5 genotype-guided dosing on clinical outcome remains to be answered, especially in the local multi-ethnic population. This pro-active approach may also sound promising for the local multi-ethnic population where majority of the renal transplant population are CYP3A5 expressers who may require a higher initial dose of FK based on genotyping profile.

ELIGIBILITY:
Inclusion Criteria:

* On follow up at SGH between the ages of 21 and 75 years old who had received or are scheduled to receive a living donor renal transplant between January 2016 to January 2023
* Has to receive tacrolimus (FK) (Prograf®; Astellas Pharma, Singapore), mycophenolic acid (MPA) (Cellcept®; Roche, Basel, Switzerland or Myfortic®; Novartis Pharma AG, Basel, Switzerland) and prednisolone as triple immunosuppressive drug maintenance regimen

Exclusion Criteria:

* Planned to be initiated on non-standard doses of tacrolimus (e.g. planned to initiate on sub-therapeutic doses of tacrolimus)
* Evidence of active liver disease or gastrointestinal disorder that might interfere with the ability to absorb oral medication
* Contraindications to tacrolimus (FK) - e.g. hypersensitivity
* Takes concurrent medications which are known to severely interact with FK (e.g. verapamil, azoles, rifampicin, erythromycin or clarithromycin

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2024-01-16 (Actual); Study Completion 2024-04-09 (Actual)

PRIMARY OUTCOMES:
Proportion of patients within the desired FK trough level at first steady state | 3 days
  E.g. Proportion of patients within target FK levels on the morning of day 3 after five unaltered FK doses
Proportion of patients within the desired FK trough level at 7 days | 7 days
  E.g. Proportion of patients within target FK levels on the morning of day 7 post initiation of FK

SECONDARY OUTCOMES:
Average FK level during the first 1 weeks after transplantation | 1 week
Average daily dose of FK the first 90 days post transplantation [days 3, 7, 14±3, 30±3, 60±3, 90±3 days post transplantation] | 90 days
Average concentration-to-dose ratio of FK during the first 90 days post transplantation [days 3, 7, 14±3, 30±3, 60+±3, 90±3 days post transplantation] | 90 days
Time to reach the first target FK range | 90 days
Number of FK dose adjustments required to reach the target FK level | 90 days
Number of markedly sub-therapeutic FK level (defined as <4 ng/mL) and markedly supra-therapeutic FK level (defined as > 20 ng/mL) | 90 days
Incidence of biopsy-proven acute rejection (BPAR), with histologic characteristics described accordingly to the Banff criteria [Banff 1997 scoring system with 2007 modifications] and/or clinically presumed acute rejection | 90 days
Incidence of graft loss (defined as failure to discontinue dialysis or if patient undergoes graft nephrectomy) | 90 days
Renal function at month 3 after transplantation. Estimated GFR (eGFR) will be calculated using CKDEPI equation. [Time Frame: at day 7, 14, 30±3, 60±3 and 90±3 days after transplantation ] | 90 days
Proportion of patients within target FK levels on day 7 post renal transplant | 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- Singapore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Shuker N, Bouamar R, van Schaik RH, Clahsen-van Groningen MC, Damman J, Baan CC, van de Wetering J, Rowshani AT, Weimar W, van Gelder T, Hesselink DA. A Randomized Controlled Trial Comparing the Efficacy of Cyp3a5 Genotype-Based With Body-Weight-Based Tacrolimus Dosing After Living Donor Kidney Transplantation. Am J Transplant. 2016 Jul;16(7):2085-96. doi: 10.1111/ajt.13691. Epub 2016 Feb 26. PMID 26714287
- [Background] Chen SY, Li JL, Meng FH, Wang XD, Liu T, Li J, Liu LS, Fu Q, Huang M, Wang CX. Individualization of tacrolimus dosage basing on cytochrome P450 3A5 polymorphism--a prospective, randomized, controlled study. Clin Transplant. 2013 May-Jun;27(3):E272-81. doi: 10.1111/ctr.12101. Epub 2013 Feb 24. PMID 23432535
- [Background] Birdwell KA, Decker B, Barbarino JM, Peterson JF, Stein CM, Sadee W, Wang D, Vinks AA, He Y, Swen JJ, Leeder JS, van Schaik R, Thummel KE, Klein TE, Caudle KE, MacPhee IA. Clinical Pharmacogenetics Implementation Consortium (CPIC) Guidelines for CYP3A5 Genotype and Tacrolimus Dosing. Clin Pharmacol Ther. 2015 Jul;98(1):19-24. doi: 10.1002/cpt.113. Epub 2015 Jun 3. PMID 25801146

DOCUMENTS (1):
  • Study Protocol (2021-09-29): https://cdn.clinicaltrials.gov/large-docs/62/NCT04825262/Prot_000.pdf